CLINICAL TRIAL: NCT04032392
Title: Immunotherapy of Advanced Hepatitis B Related Hepatocellular Carcinoma With γδT Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-013
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatitis B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous γδT cells (Experimental): Subjects will receive 3 cycles of γδT cells treatments, at four-week intervals, each cycle has 2 infusions.
  Dose escalation subjects will receive 6 infusions with dose of γδT cells escalation from 1×10e9 to 6×10e9.
  Constant dose subjects will have single infusion intravenously at a target dose of 1~2×10e9 γδT cells.
  Interventions: Biological: autologous γδT cells

INTERVENTIONS:
Biological: autologous γδT cells — Cells will be extracted by apheresis, followed by expanding and activating. The autologous γδT cells product will be adoptive transferred.

SUMMARY:
To evaluate the safety, tolerability and efficacy of autologous γδT cells in the treatment of advanced hepatitis B-related hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, open label, no control, prospective clinical trial. The study will include the following sequential phases: sign informed consent, γδT cells pre-culture, fresh biopsy and screening, apheresis, γδT cells preparation, treatment and follow-up. The study will evaluate the safety, tolerability and efficacy of autologous γδT cells in patients with advanced hepatitis B related hepatocellular carcinoma (HCC) which are refractory to current treatment.

Stage I comprising a safety cohort of patients to identify a safe dose, Stage II comprising an expanded patient group for response signal identification, Stage III to confirm efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should sign informed consent form voluntarily and comply with the requirements of this study.
2. Gender unlimited, age 18 to 70 years old.
3. Hepatocellular carcinoma histopathology proven by liver fresh biopsy.
4. According to the 2018 edition of the EASL guidelines for primary liver cancer, patients were diagnosed with advanced HBV-related hepatocellular carcinoma (BCLC stage B and C) by pathology and imaging; all patients required antiviral therapy with nucleoside analogues; other treatments (e.g. interventional therapy) at least 2 weeks prior to γδT cell infusion; patients can take the first- or second-line targeted drugs recommended by the guidelines, such as lenvatinib or sorafenib.
5. Liver function: Child-Pugh class A/B (5-9), Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
6. Expected survival ≥ 6 months.
7. Male and female of reproductive potential must agree to use birth control during the study and for at least 30 days post study.

Exclusion Criteria:

1. Combine other viral liver diseases or other liver disease patients.
2. Acute infection, gastrointestinal bleeding, etc. occurred within 30 days before screening.
3. Pregnant or lactating women; patients after organ transplantation; patients with severe autoimmune diseases; patients with uncontrolled infectious diseases.
4. Dysfunction of major organs; patient white blood cell count <1.0×10e9/L, platelet count <60×10e9/L, hemoglobin <86g/L, prothrombin time (INR) >2.3, or prolonged clotting time >6 seconds, serum albumin <28g/L, total bilirubin >51mmol/L, ALT/AST >5 times the upper limit of normal, creatinine >1.5 times the upper limit of normal.
5. Combined with other serious organic diseases, mental illnesses, including any uncontrolled clinically significant systemic diseases such as urinary, circulatory, respiratory, neurological, psychiatric, digestive, endocrine and immune diseases.
6. Allergic constitution, history of allergies to blood products, known to be allergic to test substances.
7. Immunosuppressive or systemic cytotoxic drugs may require within six months prior to screening or during treatment; 6 months prior to screening accepted other cell therapies including NK, CIK, DC, CTL and stem cell therapy etc.; immunotherapy such as PD-1 and PD-L1 antibodies.
8. Patients currently participating in other clinical trials who may violate this treatment plan and observations.
9. Those who are unable or unwilling to provide informed consent or who are unable to comply with the research requirements.
10. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed: patients with any serious acute or chronic physical or mental illness, or laboratory abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-23 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 14 months
  Incidence of adverse events (AEs) and serious adverse events (SAEs) of each patient will be recorded and analyzed.
Overall survival (OS) | 14 months
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 14 months
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the response evaluation criteria in solid tumors (RECIST) guideline.
Patients-based Quality of Life Evaluation | 14 months
  According to the European Organization for Research and Treatment of Cancer (EORTC) quality of life of the core scale criteria QLQ-C30 to evaluate and compare patients life quality before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Dr, Principal Investigator — Beijing 302 Hospital
Locations (2):
- China (2):
  - Beijing 302 Hospital of China, Beijing, Beijing Municipality
  - Beijing 302 hospital, Beijing

IPD SHARING:
Plan to Share IPD: No